CLINICAL TRIAL: NCT03573960
Title: Prospective Single Arm Post Marketing Phase IV Study to Assess the Safety and Efficacy of Lenvatinib in Subjects With Locally Recurrent or Metastatic, Progressive, Radioiodine Refractory Differentiated Thyroid Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Lenvatinib in Participants With Refractory Differentiated Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Pharmaceuticals India Pvt. Ltd (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-M091-507
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Neoplasms
Keywords: Lenvatinib, E7080, Refractory Differentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib 24 mg (Experimental): Participants will receive 24 mg (two 10-mg capsules + one 4-mg capsule) orally, once daily with or without food in 28-day cycles until disease progression or until unacceptable toxicity occurs.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules.

SUMMARY:
The purpose of this study is to evaluate the safety of lenvatinib in participants with recurrent, metastatic radio-iodine refractory differentiated thyroid cancer (DTC).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are diagnosed with locally Recurrent or Metastatic, Progressive, Radioiodine Refractory DTC, Lenvatinib naive and able to provide written informed consent.
2. Histologically or cytologically confirmed diagnosis of one of the following DTC subtypes: Papillary thyroid cancer (PTC) (including the follicular variants and other variants), Follicular thyroid cancer (FTC) (including Hurthle cell, Clear cell and Insular subtypes).
3. Measurable disease meeting the following criteria: i) At least 1 lesion >= 1.0 centimeter (cm) in the longest diameter for a non-lymph node or >= 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI). ii) Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must have shown evidence of PD based on RECIST 1.1 to be deemed a target lesion.
4. Evidence of disease progression within 12 months of screening scan.
5. Require thyroxine suppression therapy and thyroid stimulating hormone (TSH) should not be elevated (TSH should be less than [<] 4.0 milli-international units per liter [mIU/L]).
6. Participant must be radioiodine-refractory or resistant within 12 months of radioiodine therapy and have one of the following:

   * One or more measurable lesions that do not demonstrate iodine uptake on any radioiodine scan.
   * One or more measurable lesions that have substantially increased in size within 12 months of radioiodine therapy, despite demonstration of radioiodine activity at the time of that treatment by pre- or post-treatment scanning.
   * Cumulative activity of radioiodine of greater than (>) 600 milliecurie (mCi) or 22 gigabecquerels (GBq), with the last dose administered at least 6 months prior to study entry.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
8. Based on following laboratory assessment:

   * Creatinine clearance >= 30 milliliter per minute (mL/min) according to the Cockcroft and Gault formula.
   * Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to (<=) 1.5.
   * Adequate bone marrow function:

     i. Absolute neutrophil count (ANC) >=1.5*10^9/liter (L) ii. Hemoglobin >= 9.0 gram per deciliter (g/dL) (can be corrected by growth factor or transfusion) iii. Platelet count >=100 * 10^9/L
   * Adequate liver function:

     i. Bilirubin <= 1.5*upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome.

   ii. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 3*ULN (<= 5*ULN if participant has liver metastases). If ALP is > 3*ULN (in the absence of liver metastases) or > 5*ULN (in the presence of liver metastases) and participants are also known to have bone metastases, the liver-specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.
9. Urine dipstick proteinuria should be < 2+. If > or equal 2 gram (g) proteinuria is detected with dipstick, a 24-hour period urine test will be performed and the result should be < or equal to 1 g/24 hours to permit the inclusion of the patient in the clinical trial.
10. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before program entry and must agree to use a highly effective method of contraception (example, total abstinence, an intrauterine device, a double-barrier method (such as condom plus diaphragm with spermicide), a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire program.

    * If currently abstinent, participants must agree to use a double-barrier method as described above if they become sexually active during the study period or for 30 days after study drug discontinuation.
    * Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.

Exclusion Criteria:

1. Anaplastic or medullary carcinoma of the thyroid.
2. Two or more prior vascular endothelial growth factor (VEGF)/vascular endothelial growth factor receptor (VEGFR)-targeted therapies or any ongoing treatment for iodine-131 (131I) refractory DTC other than TSH-suppressive thyroid hormone therapy.
3. Blood pressure (BP) >= 140 millimeter of mercury (mmHg) Systolic and >= 90 mmHg Diastolic at screening with or without antihypertensive medications.
4. Woman who are lactating or pregnant at screening or baseline.
5. Participants who received any anticancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug. (This does not apply to the use of TSH-suppressive thyroid hormone therapy).
6. Gastrointestinal malabsorption or any other condition that in the opinion of the investigator affected the absorption of Lenvatinib.
7. Participant has history of congestive heart failure with New York Heart Association (NYHA) Classification > II, unstable angina, myocardial infarction, serious cardiac arrhythmia, or stroke within the past 6 months.
8. Electrocardiogram (ECG) with QT interval (QTc) interval >= 450 millisecond (msec). (According to Bazett's formula).
9. Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR) monitoring. (Treatment with low molecular weight heparin [LMWH] will be allowed).
10. Existing anti-cancer therapy-related toxicities of CTCAE version 4.03 grade >= 2, except alopecia and infertility.
11. Any history of or concomitant medical condition that, in the opinion of the investigator, would compromise participant's ability to safely complete the protocol.
12. Active infection (any infection requiring treatment).
13. Active malignancy (except for differentiated thyroid carcinoma, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
14. Epistaxis or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
15. Known intolerance to Lenvatinib (or any of the excipients).
16. Participants with clinically significant laboratory investigations as per the investigator's judgment.
17. Participation in any interventional clinical study within the past 90 days of enrollment to treatment.
18. Male or female of childbearing potential, unwilling to use adequate methods of contraception throughout the study.
19. Participants whom had major surgery within 3 weeks prior to study entry, or who have not recovered from prior major surgery, or whom have surgery scheduled during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Grade 2 or Higher Treatment-emergent Adverse Events | Baseline up to Week 24
  TEAEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. Adverse events (AEs) will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 where grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activity of daily living (ADL), grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL, grade 4: Life-threatening consequences; urgent intervention indicated and grade 5: Death related to AE.
Number of Dose Reductions | Baseline up to Week 24
  The number of instances of participants having to reduce the dosage of study drug based on specified toxicities.
Median Time to First Dose Reduction | Baseline up to Week 24
  Time to first dose reduction is defined as the time period from the first dose to the first dose reduction. Median time taken for the first dose reduction and 95% confidence interval will be calculated and reported.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Week 24
  ORR at 24 weeks is defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR). CR is defined as disappearance of all target and non-target lesions. All lymph nodes must be non-pathological in size (less than [<] 10 millimeter [mm] short axis). PR is defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR.
Progression-free Survival (PFS) | From date of first dose of study drug until documentation of disease progression or death from any cause (whichever occurs first) or up to approximately Week 24
  PFS is defined as the time from enrollment of participant in to study to the first sign of Progressive Disease (PD) or death due to any cause if the participant dies without experiencing PD. Disease progression per response evaluation criteria in solid tumor (RECIST) v1.1 was defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Percentage of Participants with Other TEAEs Below Grade 2 | Baseline up to Week 24
  TEAEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. The severity of all AEs will be graded according to CTCAE version 4.03 where grade 1: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Eisai Inc.
Locations (11):
- India (11):
  - Shetty's Hospital, Bangalore, Karnataka
  - Regional Cancer Centre, RCC, Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneshwar, Odisa
  - S. P. Medical College & A. G. Hospitals, Bikaner, Rajasthan
  - Tata Memorial Hospital, Mumbai
  - BL Kapoor Hospital, New Delhi, New Delhi
  - Indrayani Hospital, Alandi, Pune
  - City Cancer Centre, Vijayawada